CLINICAL TRIAL: NCT05441475
Title: A Phase 2, Open-Label Study of ABSK-011 Plus Atezolizumab to Assess Safety, Tolerability, Pharmacokinetics, and Anti-tumor Efficacy in Patients With Advanced or Unresectable Hepatocellular Carcinoma
Brief Title: A Phase 2, Open-Label Study of ABSK-011 Combined Atezolizumab in HCC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK-011-201
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Absk-011 combined with atelizumab in the treatment of patients with advanced or unresectable HCC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABSK-011 180 mg QD combined with atilizumab 1200 mg q3w. (Experimental): During part a, all subjects will receive continuous oral administration of absk-011 once a day (QD) or twice a day (bid) with an initial dose of 180 mg, and intravenous infusion (IV) of 1200 mg of atilizumab every 21 days (q3w). After the first subject (sentinel subject) in each dose cohort completed the first combined medication, follow-up subjects were administered at least 7 days later
  Interventions: Drug: ABSK-011 180 mg QD combined with atilizumab 1200 mg q3w

INTERVENTIONS:
Drug: ABSK-011 180 mg QD combined with atilizumab 1200 mg q3w — All subjects will receive continuous oral administration of absk-011 once a day (QD) or twice a day (bid) with an initial dose of 180 mg, and intravenous infusion (IV) of 1200 mg of atilizumab every 21 days (q3w).

SUMMARY:
This study is an open phase II clinical study, which consists of part a and Part B. Part a will evaluate the safety and tolerability of absk-011 combined with atilizumab in patients with advanced or unresectable HCC to And pk/pd characteristics, and determine the treatment plan of Part B. Part B will evaluate absk-011 combined with atilizumab Anti Fgf19 overexpression in advanced stage or non resectable patients who have not received systemic therapy or only received first-line systemic therapy before In addition to the safety and tolerability of HCC subjects, the antitumor activity of the combination will be further evaluated.

DETAILED DESCRIPTION:
During part a, all subjects will receive continuous oral administration of absk-011 once a day (QD) or twice a day (bid) with an initial dose of 180 mg, and intravenous infusion (IV) of 1200 mg of atilizumab every 21 days (q3w). After the first subject (sentinel subject) in each dose cohort completed the first combined medication, follow-up subjects were administered at least 7 days later.

Part B will include subjects with advanced unresectable HCC who have not previously received systemic therapy or only received first-line systemic therapy and whose Fgf19 expression is positive. No more than 70% of the enrolled subjects have only received first-line systemic therapy

ELIGIBILITY:
Inclusion Criteria:

1. before implementing any program related procedures, the subjects should understand and voluntarily sign the written informed consent and indicate the date. Subjects should be able and willing to follow the study follow-up and study procedures in the protocol.
2. there is no limit on gender, and the age when signing the informed consent is ≥ 18 years old.
3. part a: subjects with advanced or unresectable HCC who must be confirmed by histology, cytology or imaging, are not suitable for curative surgery and / or local treatment, have disease progression or cannot tolerate standard treatment after standard treatment, and have no standard treatment due to physical conditions or disease status (according to local / regional guidelines), and the child Pugh score is 5-6.

Part b: subjects with advanced or unresectable HCC who must be confirmed histologically or cytologically, are not suitable for curative surgery and / or local regional treatment, and have not previously received systematic treatment or only received first-line systematic treatment-

Exclusion Criteria:

1. history of autoimmune diseases
2. have a history of the second primary malignant tumor other than HCC within 5 years before screening,
3. have a history of uncorrectable electrolyte disorders that affect serum potassium, calcium or phosphorus levels.
4. meningeal metastasis or central nervous system (CNS) metastasis -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ABSK-011 combined with atezolizumab mab in subjects with advanced or unresectable HCC | 10 month
  Incidence of dose limiting toxicity (DLT) in the first cycle；Incidence and grade of AE, SAE and AESI by CTCAE v5.0
To evaluate the objective response rate of ABSK-011 combined with atezolizumab in subjects with advanced FGF19 overexpression or unresectable HCC | 10month
  Objective response rate (ORR): complete response and partial response determined by the investigator according to RECIST v1.1 and to be confirmed

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Hubei, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No